CLINICAL TRIAL: NCT01680393
Title: Stabilizing Cerebral and Circulatory Hemodynamics During Shoulder Surgery in the Beach Chair Position Using Sequential Compression Device (SCD) or TED Stockings Compared to a Control Group
Brief Title: Sequential Compression Device (SCD) for Stabilizing Hemodynamics in the Beach Chair Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Frank Christian Pott, MD, MD, DMSc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBH290511BRAINshoulderscd
Record Dates: First submitted 2012-02-01; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequential compression device (Experimental): During arthroscopic shoulder surgery, an SCD device will be applied to the patients legs during surgery. Cerebral oxygenation and circulatory parameters will be recorded continuously throughout the surgery. Recordings will be hidden to the primary caregiver.
  Interventions: Device: Sequential compression device
- TED stockings (Experimental): During arthroscopic shoulder surgery, TED stockings will be applied to the patients legs during surgery. Cerebral oxygenation and circulatory parameters will be recorded continuously throughout the surgery. Recordings will be hidden to the primary caregiver.
  Interventions: Other: TED stockings
- Control (No Intervention): no stockings will be applied to the patients legs

INTERVENTIONS:
Device: Sequential compression device — a sequential compression device will be applied to the legs
  Other Names: SCD express Kendall
  Arms: Sequential compression device
Other: TED stockings — TED stockings will be applied to the patients legs during surgery
  Other Names: TED compression stockings, Kendall
  Arms: TED stockings

SUMMARY:
This study is a 3-legged randomized study examining whether during shoulder surgery performed in the beach chair position active compressions of the lower leg with a sequential compression device (SCD) have a superior effect on stabilizing cerebral and circulatory hemodynamics when compared to TED stockings or a control group without any stockings.

DETAILED DESCRIPTION:
This study examines whether during shoulder surgery performed in the beach chair position active compressions of the lower leg with a sequential compression device (SCD) have a superior effect on stabilizing cerebral and circulatory hemodynamics when compared to TED stockings or a control group without any stockings.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective shoulder surgery

Exclusion Criteria:

* untreated hypertension
* no pulse in a. dorsalis pedis or a.tibialis posterior
* leg ulcers
* failed scalenous blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
cerebral oxygenation | per minute
  cerebral oxygenation averaged of 1 min during the operation

SECONDARY OUTCOMES:
ephedrine | throughout duration of anaesthesia, approximately 60 minutes
  amount of ephedrine used during surgery
cardiac output | per minute
  cardiac output averaged over 1 minute during the entire surgery
Stroke volume | per minute
  stroke volume averaged over 1 minute during the entire surgery
mean arterial pressure | per minute
  MAP averaged over 1 minute during the entire surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pott, MD,DMsc, Principal Investigator — Department of Anesthesiology, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen N, Denmark